CLINICAL TRIAL: NCT03167892
Title: Oral Screens in Post Stroke Training
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not manage to recruit enough participants
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gunilla Sandborgh Englund, professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT2017A10
Record Dates: First submitted 2017-05-11; First posted 2017-05-30 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Dysphagia, Oropharyngeal
MeSH Terms: conditions — Deglutition Disorders | interventions — Early Detection of Cancer

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Oral screen
  Interventions: Device: Oral screen
- Control (No Intervention): No intervention

INTERVENTIONS:
Device: Oral screen — Oral screen training three times per day with an effective training time of 1.5 minutes, for 3 mo
  Arms: Intervention

SUMMARY:
Stroke is a common disease in older people, and often leads to various degrees of disability. Dysphagia is one such consequence which is associated with aspiration pneumonia and malnutrition. There are studies showing that oral screen-training may reduce dysphagia, but the method is insufficiently evaluated. Since treatment with an oral screen is easy, relatively quick and cheap, it is of high relevance to perform a strict and unbiased study to assess the feasibility and efficacy of the intervention. Thus, the aim of the present study is to evaluate the effect of daily oral screen training in post-stroke patients with dysphagia.

A randomized controlled clinical study will be performed in subjects who have had a first stroke 8-12 months earlier and suffer from dysphagia. The intervention consists of daily oral screen training for 3 months. In total 70 subjects will be randomized to intervention or control. The changes in swallowing capacity is the main outcome, and secondary outcomes are subjective swallowing problems, lip force, chewing function and quality of life.

Improved oral motor function and decreased dysphagia in post-stroke patients will result in an improved quality of life for the individual, and also reduce hospitalization and health care costs.

DETAILED DESCRIPTION:
Project plan Population: Patients are recruited from the hospital Stockholms Sjukhem. When discharged, or 6-7 months after stroke, the patients are informed about the study. All positive answers are registered in a coded list. Patients are contacted by the investigators around eight months after the stroke. Patients are included in the study after informed consent, and if the inclusion criteria are fulfilled.

Inclusion criteria: ≥ 65 years of age. First stroke 8-12 months earlier. Remaining subjective and objective swallowing difficulties. Can eat. Can perform the training by himself/herself or with assistance. Natural teeth corresponding to category A according to Eichner's index.

Exclusion criteria: Moderate to severe impressive aphasia: <4.0 points by A-ning (Aphasia screening tool). Moderate to severe cognitive impairment: <23 points by MoCA (Montreal Cognitive Assessment). Unilateral neglect according to the baking tray task.

Procedure: The speech therapist screens the patient with the instruments A-ning, MoCA and Baking tray task. The dentist categorizes their dental status according to Eichner's index. Patients who do not fulfill inclusion criteria are excluded.

The patients are randomized to intervention or control group by central randomization.

At baseline, the patients in the intervention group receive an oral screen (IQoroTM) and get oral and written instructions on how to use it. They are instructed to train three times per day with an effective training time of 1.5 minutes, and to record sessions in a training diary. The patients in the control group do not get any intervention, but will be offered the corresponding training after the end of the study.

At baseline, 1.5 (intervention group only) and 3 months following intervention onset, lip force, swallowing capacity and chewing function are determined. At baseline and 3 months, oro-facial functions are screened with NOT-S and subjective swallowing problems with EAT-10 (Eating assessment tool). In order to relate these specific oral and swallowing instruments to the patient's life situation, we also include the validated instruments ESAS (Edmonton symptom assessment scale) and LiSat (Life Satisfaction) at baseline and 3 months.

Compliance in the intervention group will be evaluated by a training diary. Methods: Lip force is determined with an oral screen in the oral cavity. A hand held digital force gauge is linked to the oral screen with a wire. The patient is instructed to keep the oral screen in place as long as possible while the wire is stretched. The maximum force during tension is recorded three times.

Chewing function is evaluated with regard to bolus formation and mixing efficiency, by the use of a two-colored wax or chewing gum. The shape of the bolus and how well the colors are mixed after 30 chewing cycles is determined by visual assessment and colorimetric measures.

Swallowing capacity test (SCT) is preceded by a water swallowing test with 3-5 tea spoons of water in 4-5 rounds, in order to secure that the SCT is safe to perform. SCT: The patient is instructed to drink 150 ml of water. Swallowing speed is expressed as ml/s. Less than 10 ml/s is considered as an index of abnormal swallowing.

Power: Based on 10 ml/s as the lower limit of normal swallowing speed, we assess that 54 subjects are needed to finish the study. The estimation is made on the basis of a previous study. With 54 subjects, we will be able to determine a 40% higher proportion in the intervention group reaching 10 ml/s in SCT after finishing the training program, with 80% power and significance level 5%. To compensate for expected drop outs, we aim to recruit 35 subjects per group.

It is estimated that it will take about one year to recruit all participants to the study.

ELIGIBILITY:
Inclusion Criteria:

* First or second stroke 8-12 months earlier.
* Remaining subjective and objective swallowing difficulties.
* Can eat. Can perform the training by himself/herself or with assistance from someone.
* Natural teeth corresponding category A according to Eichner's index

Exclusion Criteria:

* Moderate to severe impressive aphasia: <4.0 points by A-ning
* Moderate to severe cognitive impairment: <23 by MoCA
* Unilateral neglect according to baking tray task

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
SCT | Change from baseline swallowing capacity baseline at 3 mo
  Swallowing capacity test

SECONDARY OUTCOMES:
Lip force | Change from baseline lip force at Month 3
  Lip muscle
Chewing function | Change from baseline bolus formation at Month 3
  Bolus formation
QoL | Change from baseline ESAS at Month 3
  Quality of Life by ESAS
Chewing function | Change from baseline mixing efficiency at Month 3
  mixing efficiency
QoL | Change from baseline LiSat at Month 3
  LiSat

CONTACTS AND LOCATIONS:
Overall Officials: Gunilla Sandborgh-Englund, Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Public Dental Service in Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appelros P, Karlsson GM, Thorwalls A, Tham K, Nydevik I. Unilateral neglect: further validation of the baking tray task. J Rehabil Med. 2004 Nov;36(6):258-61. doi: 10.1080/16501970410029852. PMID 15841602
- [Background] Bakke M, Bergendal B, McAllister A, Sjogreen L, Asten P. Development and evaluation of a comprehensive screening for orofacial dysfunction. Swed Dent J. 2007;31(2):75-84. PMID 17695052
- [Background] Bruera E, Kuehn N, Miller MJ, Selmser P, Macmillan K. The Edmonton Symptom Assessment System (ESAS): a simple method for the assessment of palliative care patients. J Palliat Care. 1991 Summer;7(2):6-9. PMID 1714502
- [Background] Fugl-Meyer AR, Melin R, Fugl-Meyer KS. Life satisfaction in 18- to 64-year-old Swedes: in relation to gender, age, partner and immigrant status. J Rehabil Med. 2002 Sep;34(5):239-46. doi: 10.1080/165019702760279242. PMID 12392240
- [Background] Hagg M, Tibbling L. Effect of oral IQoro R and palatal plate training in post-stroke, four-quadrant facial dysfunction and dysphagia: A comparison study. Acta Otolaryngol. 2015 Sep;135(9):962-8. doi: 10.3109/00016489.2015.1042043. Epub 2015 May 7. PMID 25947252
- [Background] Moller R, Safa S, Ostberg P. Validation of the Swedish translation of eating assessment tool (S-EAT-10). Acta Otolaryngol. 2016 Jul;136(7):749-53. doi: 10.3109/00016489.2016.1146411. Epub 2016 Feb 29. PMID 26924383
- [Background] Hagg M, Tibbling L. Four-quadrant facial function in dysphagic patients after stroke and in healthy controls. Neurol Res Int. 2014;2014:672685. doi: 10.1155/2014/672685. Epub 2014 Mar 4. PMID 24724023
- [Background] Schimmel M, Christou P, Miyazaki H, Halazonetis D, Herrmann FR, Muller F. A novel colourimetric technique to assess chewing function using two-coloured specimens: Validation and application. J Dent. 2015 Aug;43(8):955-64. doi: 10.1016/j.jdent.2015.06.003. Epub 2015 Jun 22. PMID 26111925
- [Background] Nathadwarawala KM, Nicklin J, Wiles CM. A timed test of swallowing capacity for neurological patients. J Neurol Neurosurg Psychiatry. 1992 Sep;55(9):822-5. doi: 10.1136/jnnp.55.9.822. PMID 1402974
- [Derived] Dalum J, Skott P, Akesson E, Persson E, Karlsson A, Habel H, Seiger A, McAllister A, Johansson K, Sandborgh-Englund G. Effect of Oral Screen Training After Stroke-A Randomised Controlled Trial. Gerodontology. 2025 Sep;42(3):380-385. doi: 10.1111/ger.12803. Epub 2024 Dec 5. PMID 39636679